CLINICAL TRIAL: NCT01274117
Title: Randomized Trial Comparing Transposition of the Basilic Vein, for Vascular Access, Performed in One-stage Versus Two-stages
Brief Title: Trial Comparing One-stage With Two-stage Basilic Vein Transposition
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PRIMARY EFFICACY OUTCOME MEASURE (MATURATION) WAS SIGNIFICANT, IN FAVOR OF THE TW0-STAGE PROCEDURE
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Stavros Kakkos, Assistant Professor, University of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2/20-4-10
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Brachiobasilic Arteriovenous Fistula
Keywords: Chronic renal failure; Basilic vein transposition fistula
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Anastomosis, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-stage transposition of the basilic vein (Placebo Comparator): One-stage transposition of the basilic vein
  Interventions: Procedure: Transposition of the basilic vein and anastomosis with the brachial vein
- Two-stage transposition of the basilic vein (Experimental): Two-stage transposition of the basilic vein
  Interventions: Procedure: Transposition of the basilic vein and anastomosis with the brachial vein

INTERVENTIONS:
Procedure: Transposition of the basilic vein and anastomosis with the brachial vein — One-stage vs two-stage transposition of the basilic vein

SUMMARY:
Arteriovenous fistulas (AVFs) are made by joining a vein to an artery in order to get the vein dilated with sufficient blood flow in order to puncture the vein and clear the blood from wastes, in patients whose kidneys are destroyed and cannot provide this function. The success rate of this procedure varies between 50-80% and depends mainly on the size of the vein, with success being higher with larger veins. One of the veins used for an AVF is the basilic vein, located at the upper arm. This vein is however deeply located and necessitates movement (transposition) during surgery to a less deep and lateral path before it is joined to the artery, in order to be used. A single study has shown that surgery performed in two parts (one to enlarge the vein and the second one to relocate the enlarged vein under the wound, not in a new path) is more successful than doing the procedure altogether.

The aim of this study is to confirm the findings of the single study mentioned above (one versus two stages of basilic vein AVF), with the difference that the vein will be relocated outside the main wound, a method that is widely accepted as being better.

DETAILED DESCRIPTION:
Arteriovenous fistulas (AVFs) are made by anastomosing a vein to an artery in order to get the vein dilated with sufficient blood flow in order to puncture the vein and perform hemodialysis in patients with renal failure. The success rate of this procedure varies between 50-80% and depends mainly on the size of the vein, with success being higher with larger veins. One of the veins used for an AVF is the basilic vein, located at the upper arm. This vein is however deeply located and necessitates transposition during surgery to a less deep and lateral subcutaneous plane before the anastomosis with the artery, in order to be used. A single study has shown that surgery performed in two stages (one to enlarge the vein and the second one to relocate the enlarged vein under the wound, not in a new path) is more successful than doing the procedure in one stage.

The aim of this study is to confirm the findings of the single study mentioned above (one versus two stages of basilic vein AVF), with the difference that the basilic vein will be relocated outside the main wound, a method that is widely accepted as being better.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure on hemodialysis
* chronic renal failure with anticipated hemodialysis

Exclusion Criteria:

* Patient unwillingness, not consenting
* Cephalic vein options
* Basilic vein less than 2.5 mm
* Basilic vein with intrinsic lesions, unsuitable for use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maturation rate | 6-10 weeks
  Usage of the AVF (or clearance in case of pre-hemodialysis)
Long term primary, primary assisted and secondary patency | 1-3 years
  Long term primary, primary assisted and secondary patency

SECONDARY OUTCOMES:
Complication rate | 1-3 years
  Hematoma, steal syndrome, venous hypertension
Basilic vein size | 4 weeks
  Basilic vein size on ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Kakkos, MD, PhD, Principal Investigator — University of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

REFERENCES:
- [Background] El Mallah S. Staged basilic vein transposition for dialysis angioaccess. Int Angiol. 1998 Jun;17(2):65-8. PMID 9754891
- [Result] Kakkos SK, Tsolakis IA, Papadoulas SI, Lampropoulos GC, Papachristou EE, Christeas NC, Goumenos D, Lazarides MK. Randomized controlled trial comparing primary and staged basilic vein transposition. Front Surg. 2015 Apr 29;2:14. doi: 10.3389/fsurg.2015.00014. eCollection 2015. PMID 25973421
- [Derived] Wang J, Gong X, Chen H, Zhong W, Chen Y, Zhou Y, Zhang W, He Y, Lou M. Causative Classification of Ischemic Stroke by the Machine Learning Algorithm Random Forests. Front Aging Neurosci. 2022 Apr 15;14:788637. doi: 10.3389/fnagi.2022.788637. eCollection 2022. PMID 35493925
- [Derived] Kaneko F, Shindo K, Yoneta M, Okawada M, Akaboshi K, Liu M. A Case Series Clinical Trial of a Novel Approach Using Augmented Reality That Inspires Self-body Cognition in Patients With Stroke: Effects on Motor Function and Resting-State Brain Functional Connectivity. Front Syst Neurosci. 2019 Dec 17;13:76. doi: 10.3389/fnsys.2019.00076. eCollection 2019. PMID 31920571
- [Derived] Battaglia G, Alesi M, Tabacchi G, Palma A, Bellafiore M. The Development of Motor and Pre-literacy Skills by a Physical Education Program in Preschool Children: A Non-randomized Pilot Trial. Front Psychol. 2019 Jan 9;9:2694. doi: 10.3389/fpsyg.2018.02694. eCollection 2018. PMID 30687164